CLINICAL TRIAL: NCT03040583
Title: Assessment of Systemic Complications (Signs) and Evolution From Patients With Sjögren's Syndrome (ASSESS)
Brief Title: The ASSESS National Multi-center Prospective Cohort
Acronym: ASSESS
Status: Recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Societe Francaise de Rhumatologie (Other)
Responsible Party: Sponsor
Other Study IDs: P060228
Record Dates: First submitted 2017-01-13; First posted 2017-02-02 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Primary Sjögren's Syndrome
Keywords: Primary Sjögren's syndrome (PSS); auto-immune diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 20 Years
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- ASSESS (PHRC) patients: Primary Sjögren's Syndrome Patients who have already participated to the study ASSESS
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — Patients data will be collected during their disease follow-up

SUMMARY:
The ASSESS national multi-center prospective cohort (Assessment of Systemic complications (Signs) and Evolution in Sjögren's Syndrome "SS") was set up in 2006 thanks to a grant of the French Ministry of Health. Fifteen centers for autoimmune diseases consecutively included consecutive patients with Primary Sjögren's Syndrome "pSS" fulfilling American-European Consensus Criteria (AECG) between 2006 and 2009. The study was approved by the Ethics Committee of Bichat Hospital in 2006. All patients gave their informed written consent. This study was followed for 5 years with the grant of the French Ministry of Health and this study will be extended for 20 years by French Society of Rheumatology (SFR). On an annual basis for a duration of 20 years, a thorough standardized paper case report form (CRF) was filled prospectively by clinicians.

DETAILED DESCRIPTION:
Primary Sjögren's syndrome (pSS) affects 0,1% of the population. This systemic autoimmune disease is characterized by disabling dryness, fatigue and pain, and systemic complications in 30% of patients. No treatment has proven effective in this disease. The previous or present systemic complications included skin, articular, lung, kidney, peripheral and central nervous system, muscular involvement and vasculitis, as well as lymphoma occurrence were recorded. For previous lymphoma, the diagnosis and the histological subtypes were confirmed by reanalysis of the medical and histological records. The objective of this cohort was to assess systemic complications (signs) and evolution of patients with pSS and to determine the evolution and factors predictors of lymphoma of systemic complications and lymphoma in pSS during a 20-years prospective follow-up. This cohort was successful in rheumatology field, 395 patients was recruited for 2 years in 15 French centers (10 rheumatology and internal medicine 5) and followed for 5 years until July 2014.

The primary objective of this cohort is to assess the evolution of Primitive Sjogren Syndrome patients and to determine predictors factors of lymphoma and systemic complications during a 20-years prospective follow-up.

ELIGIBILITY:
Inclusion Criteria:

* aged of 18 years or more
* Primary Sjögren's Syndrome Patients who have already participated to the study ASSESS

Exclusion Criteria:

* secondary Sjögren's Syndrome (SJ) associated with other autoimmune diseases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: expected population number is 395 patients
Sampling Method: Probability Sample
Enrollment: 395 (Estimated)
Dates: Start 2016-09; Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Number of patients with systemic complications during the follow-up assessed with European League Against Rheumatism (EULAR) Sjögren Syndrome Disease Activity index (ESSDAI) activity score and ESSPRI score | From the beginning of the study until the end of the 20 years follow-up
  To assess the evolution of patients with primary Sjogren's Syndrome, determine the incidence of systemic complications
Variation of complications during the follow-up assessed with ESSDAI activity score and EULAR Sjogren's Syndrome Patient Reported Index (ESSPRI) score | From the beginning of the study until the end of the 20 years follow-up
number of patient developing a lymphoma | From the beginning of the study until the end of the 20 years follow-up
  To determine the incidence of lymphomas in patients with primary Sjogren's Syndrome

SECONDARY OUTCOMES:
number of patients with cancer | From the beginning of the study until the end of the 20 years follow-up
  To analysis the incidence of cancer in patients with pSS.
number of patients with cardiovascular complication | From the beginning of the study until the end of the 20 years follow-up
  To analysis the incidence of cardiovascular complications in patients with pSS.
List of drugs taken by the patients | From the beginning of the study until the end of the 20 years follow-up
  To understand better the pathophysiology of the disease (new therapeutic targets for the pathology)
Biological report (Blood test) | From the beginning of the study until the end of the 20 years follow-up
  To Evaluate the role of biomarkers

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Mariette, Principal Investigator — SFR/AP-HP
Locations (1):
- Hopital Bicêtre, Le Kremlin-Bicêtre, Val De Marne, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Duret PM, Schleiss C, Kawka L, Meyer N, Ye T, Saraux A, Devauchelle-Pensec V, Seror R, Larroche C, Perdriger A, Sibilia J, Vallat L, Fornecker LM, Nocturne G, Mariette X, Gottenberg JE. Association Between Bruton's Tyrosine Kinase Gene Overexpression and Risk of Lymphoma in Primary Sjogren's Syndrome. Arthritis Rheumatol. 2023 Oct;75(10):1798-1811. doi: 10.1002/art.42550. Epub 2023 Jul 28. PMID 37115807